CLINICAL TRIAL: NCT00091702
Title: A Phase I/II Randomized Trial of the Safety and Immunogenicity of Cold Adapted Influenza Vaccine (FluMist) in HIV-Infected Children and Adolescents
Brief Title: Safety of and Immune Response to Two Influenza Vaccines in HIV Infected Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: P1057; 10612 (Registry Identifier: DAIDS-ES ID); PACTG P1057
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Influenza
Keywords: FluMist; Influenza Vaccine; Adolescent; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: Cold-adapted live attenuated influenza vaccine (FluMist)
Biological: Inactivated influenza vaccine (IAIV)

SUMMARY:
The purpose of this study is to compare two flu vaccines to determine their safety and ability to stimulate an immune response in HIV infected children and adolescents. This study will also determine how often and how long people who receive a vaccine are able to spread flu vaccine virus to other people.

DETAILED DESCRIPTION:
Influenza virus infections are common among children, particularly during the winter season. The infections are often mild, but more serious cases can cause a number of complications, including respiratory illnesses and bacterial infections. HIV infected children may have an increased risk for developing influenza-related bacterial complications, and influenza infections among this population may lead to more rapid disease progression. The current standard of care for HIV infected children is vaccination with an inactivated influenza vaccine (IAIV). However, IAIV is limited in its ability to stimulate the immune systems of HIV infected children with advanced disease. FluMist, a cold-adapted live attenuated influenza vaccine, is both immunogenic and effective in HIV infected children; unfortunately, FluMist is associated with viral shedding, a period of time when the influenza virus used to produce the vaccine may be transmitted to other people. This study will compare the safety and immunogenicity of IAIV and FluMist in HIV infected children and adolescents. This study will also determine the prevalence and duration of FluMist viral shedding in HIV infected children and adolescents who have received the vaccination.

Participants in this study will be randomly assigned to one of two arms. Arm A participants will receive FluMist; Arm B participants will receive IAIV. A single immunization will occur on Day 0 of the study. Arm A participants will have study visits on Days 3, 14, and 28 or home visits on Days 3 and 14. Participants in Arm B will have a study visit on Day 28. A physical exam will be performed at the initial study visit; blood will be collected at study start and at each visit thereafter. Phone calls will be made to participants throughout the study. All participants will have a final study visit after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Stable highly active antiretroviral therapy (HAART) regimen for at least 16 weeks with no changes in therapy anticipated
* Meet certain CD4 cell count and CD4% requirements
* Viral load of less than 60,000 copies/ml within 60 days prior to study start
* Received inactivated influenza vaccine (IAIV) in at least one of the past 2 years
* Written informed consent of parent or legal guardian
* Availability of parent or legal guardian to be contacted by phone

Exclusion Criteria:

* Immunosuppressive or immunomodulatory therapy within 60 days prior to immunization or immunological testing
* Aspirin or aspirin-containing therapy at the time of vaccination or planned within 42 days after immunization
* History of hypersensitivity to any component of IAIV or FluMist
* History of Guillain-Barre syndrome
* Receipt of any inactivated vaccine within 14 days prior to the study vaccination
* Receipt of any live vaccine within 30 days prior to the study vaccination
* Plans to receive any vaccine within the 30 days following the vaccination
* Receipt of any additional influenza vaccine for the duration of the study
* Prophylactic use of drugs with anti-influenza activity
* Moderate chronic pulmonary disease, obstructive or restrictive
* Cardiopulmonary disease affecting normal childhood activity
* Medically-diagnosed wheezing, bronchodilator use, or steroid use within the past 42 days
* Medical illness associated with suppression of T-cell immunity
* Pregnancy, breast-feeding, or unwillingness to use acceptable methods of contraception for 3 months following vaccination
* Severely immunosuppressed household member
* Receipt of any blood products within 3 months prior to vaccination or expected receipt during the study, including the 6-month follow-up period
* Significant fever or illness within 72 hours prior to vaccination
* Any other condition that would interfere with the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron J. Levin, MD, Study Chair — University of Colorado, Denver
Locations (61):
- United States (59):
  - UAB, Dept. of Ped., Div. of Infectious Diseases, Birmingham, Alabama
  - Univ. of South Alabama College of Medicine, Southeast Ped. ACTU, Mobile, Alabama
  - Phoenix Children's Hosp., Phoenix, Arizona
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Children's Hosp. of Orange County, Orange, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Children's Diagnostic & Treatment Ctr. of South Florida, Fort Lauderdale, Florida
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Columbus Regional HealthCare System, The Med. Ctr., Columbus, Georgia
  - Chicago Children's CRS, Chicago, Illinois
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Lawrence Family Health Ctr., Essex St. Clinic, Lawrence, Massachusetts
  - Lowell Community Health Ctr., Lowell, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Washington Univ. School of Medicine at St. Louis, St. Louis Children's Hosp., St Louis, Missouri
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Mt. Sinai School of Medicine, Div. of Ped. Infectious Diseases, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - UNC at Chapel Hill School of Medicine - Dept. of Peds., Div. of Immunology & Infectious Diseases, Chapel Hill, North Carolina
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
  - Children's Hosp. of the King's Daughters, Infectious Disease, Norfolk, Virginia
  - Seattle Children's Hospital CRS, Seattle, Washington
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Gunthard HF, Wong JK, Spina CA, Ignacio C, Kwok S, Christopherson C, Hwang J, Haubrich R, Havlir D, Richman DD. Effect of influenza vaccination on viral replication and immune response in persons infected with human immunodeficiency virus receiving potent antiretroviral therapy. J Infect Dis. 2000 Feb;181(2):522-31. doi: 10.1086/315260. PMID 10669335
- [Background] Belshe RB, Mendelman PM, Treanor J, King J, Gruber WC, Piedra P, Bernstein DI, Hayden FG, Kotloff K, Zangwill K, Iacuzio D, Wolff M. The efficacy of live attenuated, cold-adapted, trivalent, intranasal influenzavirus vaccine in children. N Engl J Med. 1998 May 14;338(20):1405-12. doi: 10.1056/NEJM199805143382002. PMID 9580647
- [Background] King JC Jr, Fast PE, Zangwill KM, Weinberg GA, Wolff M, Yan L, Newman F, Belshe RB, Kovacs A, Deville JG, Jelonek M; HIV Influenza Study Group. Safety, vaccine virus shedding and immunogenicity of trivalent, cold-adapted, live attenuated influenza vaccine administered to human immunodeficiency virus-infected and noninfected children. Pediatr Infect Dis J. 2001 Dec;20(12):1124-31. doi: 10.1097/00006454-200112000-00006. PMID 11740317
- [Background] King JC Jr, Treanor J, Fast PE, Wolff M, Yan L, Iacuzio D, Readmond B, O'Brien D, Mallon K, Highsmith WE, Lambert JS, Belshe RB. Comparison of the safety, vaccine virus shedding, and immunogenicity of influenza virus vaccine, trivalent, types A and B, live cold-adapted, administered to human immunodeficiency virus (HIV)-infected and non-HIV-infected adults. J Infect Dis. 2000 Feb;181(2):725-8. doi: 10.1086/315246. PMID 10669363
- [Result] Weinberg A, Song LY, Walker R, Allende M, Fenton T, Patterson-Bartlett J, Nachman S, Kemble G, Yi TT, Defechereux P, Wara D, Read JS, Levin M; IMPAACT P1057 Team. Anti-influenza serum and mucosal antibody responses after administration of live attenuated or inactivated influenza vaccines to HIV-infected children. J Acquir Immune Defic Syndr. 2010 Oct;55(2):189-96. doi: 10.1097/QAI.0b013e3181e46308. PMID 20581690